CLINICAL TRIAL: NCT06462404
Title: A Randomized, Double-Blind, Single-Dose, 5-Period Crossover Study to Evaluate the Efficacy, Safety, and Tolerability of E2086 Compared to Placebo and Active Comparator in Adult Subjects With Narcolepsy Type 1
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of E2086 Compared to Placebo and Active Comparator in Adult Participants With Narcolepsy Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2086-A001-101
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Narcolepsy Type 1 (NT1)
Keywords: Narcolepsy; E2086
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Sequence 1, ABECD: Placebo + E2086 Dose 1 + Active Comparator + E2086 Dose 2 + E2086 Dose 3 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 2, BCADE: E2086 Dose 1 + E2086 Dose 2 + Placebo + E2086 Dose 3 + Active Comparator (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 3, CDBEA: E2086 Dose 2 + E2086 Dose 3 + E2086 Dose 1 + Active Comparator + Placebo (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 4, DECAB: E2086 Dose 3 + Active Comparator + E2086 Dose 2 + Placebo + E2086 Dose 1 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 5, EADBC: Active Comparator + Placebo + E2086 Dose 3 + E2086 Dose 1 + E2086 Dose 2 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 6, DCEBA: E2086 Dose 3 + E2086 Dose 2 + Active Comparator + E2086 Dose 1 + Placebo (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 7, EDACB: Active Comparator + E2086 Dose 3 + Placebo + E2086 Dose 2 + E2086 Dose 1 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 8, AEBDC: Placebo + Active Comparator + E2086 Dose 1 + E2086 Dose 3 + E2086 Dose 2 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 9, BACED: E2086 Dose 1 + Placebo + E2086 Dose 2 + Active Comparator + E2086 Dose 3 (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo
- Sequence 10, CBDAE: E2086 Dose 2 + E2086 Dose 1 + E2086 Dose 3 + Placebo + Active Comparator (Experimental): Participants will receive 3 doses of E2086, an active comparator, E2086 matching placebo and active comparator matching placebo, all as oral tablets.
  Interventions: Drug: E2086; Drug: E2086 Placebo; Drug: Active Comparator; Drug: Active Comparator Placebo

INTERVENTIONS:
Drug: E2086 — E2086 oral tablets.
Drug: E2086 Placebo — E2086 matching placebo tablet.
Drug: Active Comparator — Active comparator oral tablets.
Drug: Active Comparator Placebo — Active comparator matching placebo tablet.

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of single oral doses of E2086 compared to placebo in the treatment of excessive daytime sleepiness (EDS) as assessed by the Maintenance of Wakefulness Test (MWT) in adult participants with narcolepsy type 1 (NT1).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age greater than or equal to (>=) 18 years at the time of informed consent
2. Diagnosis of NT1 defined by the following criteria:

   * History of daily periods of the irrepressible need to sleep, or daytime lapses into sleep, occurring for at least 3 months
   * History of cataplexy (which must be confirmed during the Screening Period by Sleep/Cataplexy Diary)
   * At least one of the following:

     * On Screening multiple sleep latency test (MSLT): MSL of less than or equal to (<=) 8 minutes and 2 or more sleep onset rapid eye movement periods (SOREMPs) on an MSLT performed according to standard techniques
     * On Screening nocturnal polysomnography (PSG): One or more SOREMPs within 15 minutes of sleep onset
3. Epworth Sleepiness Scale score >=10
4. Reports regular bedtime, defined as the time that the participant attempts to sleep, between 22:00 and midnight (based on data from the Screening Sleep/Cataplexy Diary)
5. Reports regular waketime, defined at the time the participant gets out of bed for the day, between 05:00 and 10:00 (based on data from the Screening Sleep/Cataplexy Diary)
6. Reports being in bed between 7 and 9 hours per night (based on data from the Screening Sleep/Cataplexy Diary)
7. Body mass index (BMI) >=18 to less than (<) 40 kilograms per meter square (kg/m^2), at Screening

Exclusion Criteria

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 international units per liter (IU/L) or equivalent units of ß-hCG [or hCG]), and females who are breastfeeding or pregnant during the Treatment Period. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the 1st dose of study drug
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

     * total abstinence (if it is their preferred and usual lifestyle)
     * a nonhormonal intrauterine device (example, "coil") or a progesterone-only intrauterine hormone-releasing system
     * a nonsteroidal oral contraceptive (participant must have been on a stable dose of the same nonsteroidal oral contraceptive product for at least 28 days before dosing and must agree to stay on the same dose of the oral contraceptive throughout the study and for 28 days after study drug discontinuation.)
     * depot medroxyprogesterone acetate or depot norethisterone enantate.
     * have a vasectomized partner with confirmed azoospermia.
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 30 days after study drug administration.

     * Participants on an oral contraceptive must use an additional barrier method throughout the study and for 30 days after study drug administration.

   NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that are, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
3. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners meet the exclusion criteria above that is, the female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period and for 92 days after study drug administration. No sperm donation is allowed during the study period and for 92 days after study drug administration
4. History of myocardial infarction, ischemic heart disease, or cardiac failure at Screening
5. History of clinically significant arrhythmia or uncontrolled arrhythmia
6. Known to have or probable positivity for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within 14 days of any study visit.
7. Exposure within the last 10 days to an individual with confirmed or probable coronavirus disease-2019 (COVID-19) or symptoms within the last 10 days that are on the most recent Centers for Disease Control and Prevention (CDC) list of COVID symptoms
8. Hypersensitivity to excipients of the study drug (E2086), or to active comparator or any of its excipients
9. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the CSSRS)
10. Any lifetime suicidal behavior (per the Suicidal Behavior section of the C-SSRS)
11. Any history of psychiatric disease (including but not limited to depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, anxiety disorders), within 10 years of Screening
12. Any current psychiatric symptoms as indicated by a standard screening tool (Diagnostic and Statistical Manual of Mental Disorders [DSM-5] Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult)
13. Participants with one or more 1st degree (blood) relatives who have lifetime diagnosis of bipolar type I disorder or a psychotic disorder
14. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics within 2 years before Screening
15. Evidence of clinically significant disease (examples, allergies; cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
16. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline
17. Any history of or concomitant medical condition that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study.
18. History of drug or alcohol dependency or abuse within 2 years before Screening
19. Use of illegal recreational drugs at Screening and throughout the study
20. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
21. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5* the half-life, (whichever is longer) preceding informed consent.
22. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing (examples, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system)
23. History of formally diagnosed moderate to severe obstructive sleep apnea, current use of continuous positive airway pressure, or symptomatic restless legs syndrome
24. Apnea-hypopnea index >=15 on Screening PSG
25. Periodic limb movement arousal index (PLMAI)>=15 on Screening PSG
26. Use of anti-cataplectic medications within 5* the half-life before Screening
27. Use of psychostimulant medications, prescription and over-the-counter (OTC), within 5*the half-life before Screening

    - Examples of prohibited medications include OTC stimulants (example, pseudoephedrine), methylphenidate, amphetamines, modafinil, armodafinil, sodium oxybate, and pemoline
28. Use of sleep promoting medications, prescription and OTC, within 28 days or 5*the half-life before Screening - Examples of prohibited medication include OTC sleep aids, trazodone, hypnotics, benzodiazepines, barbiturates, cannabinoids, and opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Mean Sleep Latency (MSL) as Assessed by the 4 Maintenance of Wakefulness Tests (MWTs) for E2086 Versus Placebo at Day 1 | At Day 1
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of excessive daytime sleepiness (EDS) which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.
MSL as Assessed by the 4 MWTs for E2086 Versus Placebo at Day 5 | At Day 5
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of EDS which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.
MSL as Assessed by the 4 MWTs for E2086 Versus Placebo at Day 9 | At Day 9
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of EDS which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.
MSL as Assessed by the 4 MWTs for E2086 Versus Placebo at Day 13 | At Day 13
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of EDS which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.
MSL as Assessed by the 4 MWTs for E2086 Versus Placebo at Day 17 | At Day 17
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of EDS which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.

SECONDARY OUTCOMES:
MSL as Assessed by the 4 MWTs for E2086 Versus Active Comparator | Days 1, 5, 9, 13 and 17
  Sleep latency is defined as the amount of time a person takes to fall asleep. The MWT is an objective assessment of EDS which consists of measurement tests. A participant undergoes four 40-minute wake trials, where an increased ability to stay awake in the context of trying to remain awake is reflected in a prolonged sleep latency. These measurements of sleep latency at regular intervals across the day are averaged to calculate the mean sleep latency. The MWT will be performed as per the 2021 guidance of the American Academy of Sleep Medicine.
Karolinska Sleepiness Scale (KSS) Score for E2086 Versus Active Comparator | Day 1 up to Day 18
  The KSS is a subjective measure of an individual's level of sleepiness during the last 10 minutes, as assessed at a particular time of day. The KSS is rated on a 10-point scale, from 1 = extremely alert, to 10 = extremely sleepy, falls asleep all the time. Higher score indicates more sleepiness.
KSS Score for E2086 Versus Placebo | Day 1 up to Day 18
  The KSS is a subjective measure of an individual's level of sleepiness during the last 10 minutes, as assessed at a particular time of day. The KSS is rated on a 10-point scale, from 1 = extremely alert, to 10 = extremely sleepy, falls asleep all the time. Higher score indicates more sleepiness.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first dose of study drug up to Day 20
Number of Participants With Markedly Abnormal Clinical Laboratory Values | Baseline up to Day 20
  Clinical laboratory will include hematology, chemistry, and urinalysis.
Number of Participants With Markedly Abnormal Vital Sign Values | Baseline up to Day 20
  Vital sign parameters will include systolic and diastolic blood pressure, pulse, respiratory rate, body temperature.
Number of Participants With Markedly Abnormal Electrocardiogram (ECGs) Findings | Baseline up to Day 20
Number of Participants With Markedly Abnormal Electroencephalogram (EEGs) Findings | Baseline up to Day 20
Number of Participants With Suicidality as Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS) | Baseline up to Day 20
  Suicidality will be assessed using the C-SSRS. The C-SSRS assesses an individual's degree of suicidality, including suicidal ideation and suicidal behavior. The C-SSRS is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior is indicated when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation is indicated when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Cmax: Maximum Observed Plasma Concentration of E2086 and its Metabolite M1 | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
Tmax: Time to Reach Cmax of E2086 and its Metabolite M1 | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration of E2086 and its Metabolite M1 | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Zero Time Extrapolated to Infinite of E2086 and its Metabolite M1 | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
t½: Terminal Phase Half-life of E2086 and its Metabolite M1 | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
MRp: Metabolite Ratio of AUC(0-inf) | Days 1, 5, 9, 13 and 17: 0-24 hours post-dose
  MRp will be calculated as ratio of plasma AUC(0-inf) of metabolite to parent following molar correction.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - SDS Clinical Trials, Santa Ana, California
  - PharmaDev Clinical Research, Miami, Florida
  - Sleep Practioners, LLC, Macon, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Sound Asleep Research, Inc., Lansing, Michigan
  - Research Carolina Elite, Denver, North Carolina
  - Medical Care Inc., Goldsboro, North Carolina
  - Advances Repiratory and Sleep Medicine, Greensboro, North Carolina
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
- Canada (2):
  - AMDX Inc., Markham, Ontario
  - Jodha Tishon Inc, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.